CLINICAL TRIAL: NCT05972642
Title: A Prospective, Single Center, Single Group, Pivotal Clinical Trial to Evaluate the Safety and Efficacy of Non-Invasive Procedures Using Ultrasound-Guided High-Intensity Focused Ultrasound 'Sonotrip V20'
Brief Title: Safety & Efficacy of Non-Invasive Procedures Using Ultrasound-Guided HIFU 'Sonotrip V20' in Symptomatic Uterine Fibroids
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Jeysis Medical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU-PCT
Record Dates: First submitted 2023-06-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Myoma;Uterus
Keywords: Ultrasound-guided HIFU; Symptomatic uterine fibroids; Safety and efficacy; Sonotrip V20
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Intervention Model Description: This is a single-arm study.
Masking Description: As this is a single-arm study, there will be no separate randomization and blinding procedures. However, to minimize bias to the efficacy assessor, an imaging assessor independent of the investigator will be assigned to assess the percentage reduction in uterine fibroid volume.
  The independent assessor will use MR imaging to assess the volume of the uterine fibroids at screening versus the volume of the uterine fibroids at 24 weeks post-procedure and the volume of the nonperfused area immediately post-procedure. In addition, the independent assessor's assessment notes will be kept secure for the duration of the study and will not be accessible to anyone other than the independent assessor. Once all assessments are completed for a subject, they will be forwarded to the Data Controller in batches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU treatment (Experimental): Eligible patients will be treated with HIFU instrument.
  Interventions: Device: HIFU-treatment

INTERVENTIONS:
Device: HIFU-treatment — The investigator will sedate the subject and perform the HIFU procedure with the investigational medical device according to the pre-established procedure plan (see Table 11 for procedure plan) (procedure may take up to 2 hours). During the procedure, the investigator may modify the pre-established procedure plan by checking in with the subject occasionally to assess the presence of heat and pain at the site of the investigational device application.
  Other Names: Treatment arm

SUMMARY:
This is a single-arm clinical trial evaluating the safety and efficacy of ultrasound-guided HIFU (Sonotrip V20) for symptomatic uterine fibroids. 57 cases will be enrolled at a Korean institution. Participants will undergo the HIFU procedure based on a pre-established plan using MRI images. Assessments will be conducted immediately post-procedure and at 4 and 24 weeks. Primary endpoint is fibroid volume reduction at 24 weeks, with secondary endpoints including Non-Perfused Volume Ratio, quality of life, hemoglobin change, pain assessment, and additional medication use. Adverse events will be monitored.

DETAILED DESCRIPTION:
This study is designed as a prospective, single-center, single-arm, confirmatory clinical trial to evaluate the safety and efficacy of the ultrasound-guided High-Intensity Focused Ultrasound (HIFU) device 'Sonotrip V20' in patients with symptomatic uterine fibroids, and includes a total of 57 cases (considering a dropout rate of 20%) at one institution in Korea.

After receiving a full explanation of the study, volunteers who voluntarily agree in writing to participate in this study and are found to meet the inclusion/exclusion criteria will be enrolled in the study, assigned a subject registration number, and scheduled for hospitalization and procedure. The investigator will develop a procedure plan from the MRI images prior to the procedure date and perform the HIFU procedure according to the pre-established procedure plan on the day of the procedure.

Subjects will undergo observations and tests (such as pregnancy tests and laboratory tests) to evaluate efficacy and safety immediately after the procedure and at 4 and 24 weeks after the procedure.

The primary efficacy endpoint to evaluate the safety and efficacy of the investigational medical device is "reduction in uterine fibroid volume (%) at 24 weeks post-procedure," and the secondary efficacy endpoints are "Non-Perfused Volume Ratio (NPVR) immediately after the procedure," "quality of life (score)," "post-procedure hemoglobin change (%)," "pain assessment during the procedure (score)," and "percentage of subjects receiving additional sedation or pain medication (N%). Safety is assessed by the number of adverse events that occurred in subjects during the study.

ELIGIBILITY:
Inclusion Criteria:

1. adult women 19 years of age or older
2. with symptomatic uterine fibroids* (e.g., heavy periods, dysmenorrhea, abnormal bleeding, pressure symptoms including pelvic pain, and urinary and bowel dysfunction)12

   *Symptomatic fibroids: a Symptom Severity Score (SSS) score of 41 or higher on the UFS-QOL questionnaire for fibroid symptoms.
3. premenopausal (FSH<40 mIU/ml)
4. For women of childbearing potential, agree to use at least one clinically adequate method of contraception* for the duration of the study.

   * Clinically adequate contraception is defined as "[intrauterine device (e.g., Loop, Mirena), chemical barrier method (spermicide), or subdermal implant (e.g., Implanon)] + physical barrier method (male or female)", tubal surgery, or laparoscopic contraception (a type of tubal ligation).
5. have been diagnosed with fibroids by imaging studies.
6. have four or fewer fibroids to be treated
7. the size of the fibroids to be treated is 12 cm or less with no necrotic or calcified areas13
8. have voluntarily decided to participate in this study and have given written consent to the informed consent form and the study protocol
9. willing to comply with the protocol

Exclusion Criteria:

1. suspected intrauterine malignancy on contrast MR scan (however, if endometrial biopsy confirms that the lesion is not malignant, the patient may be eligible to participate in the study)14, 15, 16
2. the lesion to be treated is adenomyosis or highly perfused fibroid*17

   *highly perfused fibroid is defined as having an image intensity equal to or greater than the myometrium on T2-weighted images.
3. Planning to become pregnant in the future, or currently pregnant (women of childbearing potential who are β-hCG positive are not eligible to participate in the study).
4. Have a contraindication to MRI examination (e.g., claustrophobia) or a history of hypersensitivity to gadolinium-based contrast agents (MR contrast agents) or ultrasound contrast agents However, if any of the above can be controlled with medication, patients may be eligible to participate in the study.
5. currently being treated with or having been treated with gonadotropin-releasing hormone agonists (GnRHa) (however, if 12 weeks have elapsed since the end of GnRHa treatment, patients may participate in the study)
6. the fibroids to be treated are not measurable on MRI
7. the location of the fibroids to be treated falls into type 7 and/or type 8 according to the following classification

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Volume reduction | An independent imaging assessor will calculate the uterine fibroid volume on MR images taken at screening and 24 weeks post-procedure to assess the percentage reduction in uterine fibroid volume from screening to 24 weeks post-procedure.
  Uterine fibroid volume reduction at 24 weeks post-procedure (%)

SECONDARY OUTCOMES:
NPVR | within 24 hours of the procedure
  An independent imaging assessor will evaluate the ratio of the volume of the uterine fibroids at screening to the volume of the nonperfused area immediately after the procedure (within 24 hours of the procedure) using MR imaging. Percentage of the volume of non-perfused tissue (tissue that is not enhanced on contrast MR imaging because it is necrotic and not flowing with blood from the HIFU procedure) by volume of uterine fibroids.
Quality of life-SF36 | Evaluate changes in quality of life before and after 4 weeks and 24 weeks after procedure
  It is a questionnaire for assessing overall quality of life and consists of 36 questions in eight domains: physical functioning, role limitation-physical, bodily pain, general health, vitality, social functioning, role limitation-emotional, mental health, and other health status change questions.
Quality of life-UFS-QOL | Evaluate changes in quality of life before and after 4 weeks and 24 weeks after procedure
  This questionnaire is designed to assess quality of life related to uterine fibroid symptoms and consists of an 8-item Symptom Severity Score and a 29-item Quality of Life Questionnaire.
Hct change | Evaluate the rate of change in hemoglobin (Hb) from pre-procedure to 4 and 24 weeks post-procedure.
  Post-procedure hemoglobin change (%)
Intra-procedural pain assessment | During the time of procedure
  After the procedure, a self-completed Numerical Rating Scale (NRS), 0-10 questionnaire will be used to assess pain from the HIFU procedure during the procedure.
Percentage of subjects who received additional sedation or pain medication (N%) | During and after the procedure within 24 hours
  Evaluate the percentage of subjects who received additional sedation or analgesia during the procedure and within 24 hours after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, Principal Investigator — Seoul National University Hospital